CLINICAL TRIAL: NCT01710800
Title: Twenty-Four Hour Combined Multi-Channel Impedance and pH Ambulatory Monitoring: Impedance Reflux Episodes of Patients On and Off Proton Pump Inhibitor Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Fouad Moawad, Gastroenterologist, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 20593-8
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2012-11

CONDITIONS: GERD
Keywords: impedance; reflux; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo arm (Placebo Comparator): Patients will be randomized to receive either PPI or placebo and then undergo a 24 hour pH study with impedance to measure the number of reflux episodes
  Interventions: Drug: placebo
- Esomeprazole (Active Comparator): Patients were randomly assigned to receive 40 mg esomeprazole twice daily prior to undergoing a 24 hour pH study with impedance to measure the number of reflux episodes
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole
  Other Names: Nexium
  Arms: Esomeprazole
Drug: placebo
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to determine the effects of proton pump inhibitors (PPIs) on the total number of reflux episodes in the distal esophagus measured by impedance in patients with and without gastroesophageal reflux disease (GERD) based on 24-hour pH testing. In addition to changing the acidity of the refluxate, the investigators hypothesize that PPIs also reduce the total number of reflux episodes due to its anti-secretory effects.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients (age 18 or older) with reflux symptoms willing to participate

Exclusion Criteria:

* Pregnancy
* Prior esophageal or gastric surgery
* Achalasia
* Scleroderma
* Gastroparesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

REFERENCES:
- [Derived] Moawad FJ, Betteridge JD, Boger JA, Cheng FK, Belle LS, Chen YJ, Maydonovitch CL, Wong RK. Reflux episodes detected by impedance in patients on and off esomeprazole: a randomised double-blinded placebo-controlled crossover study. Aliment Pharmacol Ther. 2013 May;37(10):1011-8. doi: 10.1111/apt.12301. Epub 2013 Apr 7. PMID 23560727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible patients with suspected GERD will be referred to the manometry and reflux lab testing for potential recruitment into the study
Pre-assignment Details: Prior to undergoing 24 hour pH with impedance, all participants will receive either one week of esomeprazole or one week of placebo.
Groups:
- First Intervention (7 Days), Second Intervention (7 Days): Patients will be randomized to receive either PPI or placebo (sequence 1) for 7 days and then undergo a 24 hour pH study with impedance to measure the number of reflux episode. The second sequence of medications (that is either placebo or PPI or sequence 2) will be administered followed by repeat 24 hour pH with impedance 7 days later.
Period: Overall Study
Arm/Group | First Intervention (7 Days), Second Intervention (7 Days)
Started | 63 (63 patients consented to be part of the study)
Received PPI Intervention | 44
Received Placebo Intervention | 45
Completed | 41 (22 drop outs(consented but did not participate, refused 2nd intervention))
Not Completed | 22
Not completed — Withdrawal by Subject | 21
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients will be randomized to receive either PPI or placebo (sequence 1) and then undergo a 24 hour pH study with impedance to measure the number of reflux episodes. Sequence 2 (placebo or PPI) will be administered followed by repeat 24 hour pH with impedance.
Arm/Group | All Study Participants
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Impedance Episodes Following PPI and Placebo
Description: Impedance is defined as a 50% decrease from baseline in retrograde movement of liquid from the stomach to the esophagus. In other words, it measures the number of retrograde reflux episodes.
Time Frame: 1 week
Population: We analyzed as per protocol. Only patients who completed both 24 hour pH studies with impedance were analyzed.
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Placebo Arm | Esomeprazole
Number analyzed (Participants) | 41 | 41
number of episodes | 47 (22) | 53 (29)

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Placebo Arm | PPI Arm
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44

LIMITATIONS AND CAVEATS:
Single center study. Relatively small number of patients studied, although recruitment goal reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No